CLINICAL TRIAL: NCT05117515
Title: Retrospective Monocentric, Observational PMCF - Study on the Performance and Safety of Uni-Graft® K DV Patch in Patients With Vascular Reconstructions
Brief Title: Retrospective Study of the Uni-Graft® K DV Patch in the Clinical Routine
Acronym: RESTUGPA
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2116
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Femoral Artery Stenosis; Iliac Artery Stenosis; Carotid Artery Stenosis
Keywords: Reconstructive interventions; vascular patch; polyethylene terephthalate
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uni-Graft KDV Patch
  Interventions: Device: Vascular reconstruction

INTERVENTIONS:
Device: Vascular reconstruction — Vascular reconstructions in the carotid, profunda, femoral and iliac arteries

SUMMARY:
Uni-Graft® K DV Patch is marketed in Europe since 1999 for reconstructive interventions of the deep femoral, femoral and iliac artery and was also indicated for carotid interventions until 01/2020. Previous studies focused on the clinical performance of different patch materials used for patch angioplasty in different indications, without specifying the product or manufacturer. Thus, it is not surprising that there is a limited amount of published literature available describing the use of the Uni-Graft® K DV Patch in the clinical routine. Therefore, the aim of the present non-interventional study (NIS) is to close this gap by collecting and evaluating existing safety and performance data documented in the clinical routine especially during the application of the Uni-Graft® K DV Patch.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* written informed consent
* treated with Uni-Graft® K DV Patch for reconstructive interventions of the carotid, deep femoral, femoral and iliac artery

Exclusion Criteria:

* Use of the Uni-Graft® K DV Patch if allergies to components of the patch are known
* Use of the Uni-Graft® K DV Patch in case of a known hypersensitive reaction to the patch and / or its components (e.g. polyethylene terephthalate).
* No use of Uni-Graft® K DV Patch
* Use of Uni-Graft® K DV Patch outside the intended use of the product at the date of application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients with an age ≥ 18 years at intervention, who had provided written informed consent and had been treated with Uni-Graft® K DV Patch will be eligible for documentation in this NIS. Patients who had received Uni-Graft® K DV Patch not for reconstructive interventions of the carotid, deep femoral, femoral and iliac artery will be not included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Restenosis Rate in postoperative Course | approximately up to 3 months after Implantation
  Retrospective evaluation of restenosis rate from information documented in the patient file: the NASCET is an angiographic measurement recommended by the "North American Symptomatic Carotid Endarterectomy Trial"-Group. According to the NASCET-Method the grade of stenosis in relation to the diameter of the ACI distal to the stenosis in the area of the parallel arterial wall is measured.

SECONDARY OUTCOMES:
Postoperative bleeding | approximately up to 3 months after Implantation
  Retrospective evaluation of restenosis rate from information documented in the patient file: Report of any bleeding during postoperative course
Rate of Intraoperative stroke | intraoperatively
  Retrospective evaluation of stroke rate from information documented in the patient file: Report of any intraoperative stroke
Rate of postoperative stroke | approximately up to 3 months after Implantation
  Retrospective evaluation of stroke rate from information documented in the patient file: Report of any stroke during postoperative course
Rate of patch related infections | approximately up to 3 months after Implantation
  Retrospective evaluation of any patch related infections from information documented in the patient file: Report of any patch related infections during postoperative course
Rate of postoperative nerve lesions | approximately up to 3 months after Implantation
  Retrospective evaluation of nerve lesion rate from information documented in the patient file: Report of any postoperative nerve lesions postoperative course
Rate of postoperative pseudoaneurysm | approximately up to 3 months after Implantation
  Retrospective evaluation of pseudoaneurysm rate from information documented in the patient file: Report of any postoperative pseudoaneurysm during postoperative course
Primary and secondary patency rate | approximately up to 3 months after Implantation
  Retrospective evaluation of primary and secondary patency rate from information documented in the patient file during postoperative course
Freedom of re-intervention rate | approximately up to 3 months after Implantation
  Retrospective evaluation of re-intervention rate from information documented in the patient file: Report of any re-intervention during postoperative course

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany